CLINICAL TRIAL: NCT03141710
Title: Effect of Prebiotic in Type 2 Diabetes (Diabetes and Health Study)
Brief Title: Commercial Prebiotic Supplement Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Study 805
Record Dates: First submitted 2017-02-08; First posted 2017-05-05 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: 20ml of prebiotic per day for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12 type 2 diabetes patients (Experimental): Long-term dietary (12 weeks) intervention of 20ml of prebiotic per day
  Interventions: Dietary Supplement: 20 ml of prebiotic per day

INTERVENTIONS:
Dietary Supplement: 20 ml of prebiotic per day — 12 volunteers will take 20ml of prebiotic per day for 12 weeks

SUMMARY:
Previous work in 2015/16 has identified changes in the gut microbiota with prebiotic (Molkosan®) supplement. It report significant changes in metabolic health bio-markers and faecal SCFA profile in 18 health adult subjects consuming 20 ml of product twice a day. Improvement in fasting metabolic parameters was observed flowing the intervention period. A reduction on Total Cholesterol, Glucose, Triglycerides and Insulin was observed.

In this study, a lower dose (20ml/d) in subjects with type 2 diabetes will be examed, over an extended period of time (12 week period) to match the profile of the intended consumer and provide preliminary data to support a larger multi-centre trial.

DETAILED DESCRIPTION:
The study will be conducted in males and females with type 2 diabetes managed by diet and lifestyle alone.

The participants who meet the inclusion and exclusion criteria of the study will attend a screening visit where they will complete a medical screening and sign the consent form for participation in the study. Participates will visit the Human Nutrition Unit at the Rowett Institute to provide samples at week 0 (baseline), week 6 and week 12.

Participants' height, weight, and blood pressure will also be recorded. The investigators will measure HbA1c by a finger prick blood sample to confirm whether participants are a prediabetic or type 2 diabetic subjects. A 3-day weighed intake food diary will be completed during the initial washout period (minimum of 7 days) of the study in order to note their normal eating habits. No probiotic or prebiotics to be consumed during washout period and study period.

During the study periods, participants will take 20ml of prebiotic daily over the 12 consecutive weeks.

For the study visits, each participant will undergo, on two separated occasions, an OGTT, with and without the product at week 0 (to assess acute effects, prior to chronic ingestion) and at week 12 (to assess acute effects after chronic ingestion). The two OGTTs (with and without test product) will be separated by a period of 48 hr. Thus, each participant will have four OGTTs during the study. To minimise systematic errors, one half of the participants will start with the test product OGTT and the other half will start without product OGTT. The starting order will be determined randomly. Six blood samples will be collected during the course of 3 hours (0, 30, 60, 90,120 and 180 min) using a cannulation after consuming 75 g of Polycal liquid (glucose load). Together with OGTT, breath samples will be taken every 30 min for measuring hydrogen and methane.

Only one fasted blood sample will be taken at week 6 (OGTT will not be performed at week 6).

Finger prick blood sample will be taken at week 12 to monitor for changes in HbA1c levels after prebiotic supplement.

Plasma samples will be collected from all blood samples from OGTTs and week 6 blood sample. Plasma glucose and lipid profiles (total cholesterol, HDL, LDL and triglycerides) will be measured by KONI analysis at the University of Aberdeen. Insulin will be measured by ELISA by researchers. All the plasma samples which are taken before and after taking the prebiotic supplement also be analysed for GLP-1, GIP, c-peptide and glucagon analysis by luminex assay.

GLP-1 and GIP are incretins which are produced in the intestinal mucosa and are normally secreted when food is eaten in order to reduce glycaemic exclusion by causing an increase in insulin secretion. These incretins are involved in the early stage of the insulin secretory response however the plasma insulin response is also influenced by hepatic insulin extraction which GLP-1 and GIP measurement cannot determine, therefore to optimise this, C-peptide will be also measured in this study.

All the data will be compared before and after supplementation and values are presented by means ± standard deviations.

From the faecal samples, the SCFA content of the samples to be determined by capillary gas chromatography. SCFA to be quantified against authentic standards of acetate, propionate, butyrate, valerate and the branched chain fatty acids iso-butyrate and iso-valerate. The lower limit for reliable detection of each product is 0.2 mM. DNA to be extracted at University of Aberdeen using the FastDNA spin kit for faeces following the manufacturer's instructions and quantitative PCR (qPCR). Samples and standards are prepared in 96 well plate format, enabling the use of a multichannel pipettes for setting up the running plate. PCR primer sets and amplification conditions are as described in previous studies.

The complete dataset will be analysed and values will be presented as a mean value and standard deviation. Then the baseline value and the value after supplementation (at 6 and 12 weeks) will be compared. Statistically significantly differences will be calculated by statistician with power calculate.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance (IGT, identified by HbA1c) or type 2 diabetes (lifestyle management; identified by HbA1c) age 18-65, with BMI 18-40 kg m-2, measured at screening visit.

Exclusion Criteria:

* Type 1 Diabetes, Severe gastrointestinal disorders (IBD), Kidney disease, Thromboembolic or coagulation disease, Hepatic disease, Alcohol or any other substance abuse, Eating disorders, Unregulated thyroid disease, Antibiotic use within the last 3 months, including proscribed and prescribed use. Current probiotic use or prebiotic use. Medication for glucose regulation. Female with breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change of oral glucose tolerance test (OGTT) | At baseline and 12 weeks prebiotic consumption
  Six blood samples will be collected during the course of 3 hours (0, 30, 60, 90,120 and 180 min) using a cannulation after consuming 75 g of Polycal liquid (glucose load). Plasma glucose level will be measured by KONI analysis and

SECONDARY OUTCOMES:
Change of insulin levels | At baseline, 6 weeks and 12 weeks prebiotic consumption
  Six blood samples will be collected during the course of 3 hours (0, 30, 60, 90,120 and 180 min) using a cannulation after consuming 75 g of Polycal liquid (glucose load). insulin level will be measured by luminex assay.
HbA1c measured by Alere Afinion™ AS100 Analyzer | At baseline and 12 weeks prebiotic consumption
  The term HbA1c refers to glycated haemoglobin. It develops when haemoglobin, a protein within red blood cells that carries oxygen throughout the body. By measuring glycated haemoglobin (HbA1c) can indicate blood sugar levels.
  Finger prick method will be introduced to collect the small amount of blood samples into the Alere Afinion™ AS100 Analyzer cartridge. Insert cartridge to the machine to read the data. Inclusion criteria will be the levels above 6 % (42mmol/mol). We will also measure HbA1c at 12 week to monitor for changes.
Change of BMI (kg/m^2) measurement | At baseline and 12 weeks prebiotic consumption
  Weight or Body Mass is defined as the quantity of matter in the body, measured by weight (kg) i.e. the force that matter exerts under standard gravitational effect. Height (m) will be recorded for conjunction with weight measurements to calculate Body Mass Index (BMI) values.
Change of Total Cholesterol levels | At baseline, 6 weeks and 12 weeks prebiotic consumption
  Total cholesterol (HDL and LDL -Cholesterols) will be measured by KONI analysis at University of Aberdeen. Separately measured HDL- and LDL-cholesterols levels will be combined for total cholesterol levels.
Change of GLP-1 levels | At baseline, 6 weeks and 12 weeks prebiotic consumption
  The incretin hormones, glucagon-like peptide-1 (GLP-1) secretion, contributes to glucose intolerance. GLP-1 levels will be measured by luminex assay.
Change of GIP levels | At baseline, 6 weeks and 12 weeks prebiotic consumption
  Glucose-dependent insulinotropic polypeptide (GIP) is potentiate the insulin response to nutrients. Insulinotropic capacity of GIP is markedly diminished in type 2 diabetes. Incretin hormone GIP will be measured by luminex assay.
Change of triglyceride levels | At baseline, 6 weeks and 12 weeks prebiotic consumption
  Triglyceride levels will be measured for identifying the lipid profiles. Triglyceride will be measured by KONI analysis.
Change of C-peptide levels | At baseline, 6 weeks and 12 weeks prebiotic consumption
  C-peptide are involved to hepatic insulin extraction. C-peptide levels are measured by luminex assay.
Change of glucagon levels | At baseline, 6 weeks and 12 weeks prebiotic consumption
  Glucagon levels will be measured by luminex assay.
Change of fermentation markers | At baseline and 12 weeks prebiotic consumption
  Breath samples will be measured hydrogen and methane levels

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M Johnstone, PhD, Principal Investigator — University of Aberdeen, The Rowett Institute
Locations (1):
- The Rowett Institute, Human Nutrition Unit, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson GR, Roberfroid MB. Dietary modulation of the human colonic microbiota: introducing the concept of prebiotics. J Nutr. 1995 Jun;125(6):1401-12. doi: 10.1093/jn/125.6.1401. PMID 7782892
- [Background] Kenteu B, Noubiap JJ, Etoa MC, Azabji-Kenfack M, Dehayem M, Sobngwi E. Acute glycaemic effects of co-trimoxazole at prophylactic dose in healthy adults. BMC Endocr Disord. 2016 Nov 15;16(1):62. doi: 10.1186/s12902-016-0142-6. PMID 27927207
- [Background] Marathe CS, Rayner CK, Lange K, Bound M, Wishart J, Jones KL, Kahn SE, Horowitz M. Relationships of the early insulin secretory response and oral disposition index with gastric emptying in subjects with normal glucose tolerance. Physiol Rep. 2017 Feb;5(4):e13122. doi: 10.14814/phy2.13122. Epub 2017 Feb 27. PMID 28242817
- [Background] Salonen A, Lahti L, Salojarvi J, Holtrop G, Korpela K, Duncan SH, Date P, Farquharson F, Johnstone AM, Lobley GE, Louis P, Flint HJ, de Vos WM. Impact of diet and individual variation on intestinal microbiota composition and fermentation products in obese men. ISME J. 2014 Nov;8(11):2218-30. doi: 10.1038/ismej.2014.63. Epub 2014 Apr 24. PMID 24763370
- [Background] Walker AW, Ince J, Duncan SH, Webster LM, Holtrop G, Ze X, Brown D, Stares MD, Scott P, Bergerat A, Louis P, McIntosh F, Johnstone AM, Lobley GE, Parkhill J, Flint HJ. Dominant and diet-responsive groups of bacteria within the human colonic microbiota. ISME J. 2011 Feb;5(2):220-30. doi: 10.1038/ismej.2010.118. Epub 2010 Aug 5. PMID 20686513
- [Background] Yanagimachi T, Fujita Y, Takeda Y, Honjo J, Sakagami H, Kitsunai H, Takiyama Y, Abiko A, Makino Y, Kieffer TJ, Haneda M. Dipeptidyl peptidase-4 inhibitor treatment induces a greater increase in plasma levels of bioactive GIP than GLP-1 in non-diabetic subjects. Mol Metab. 2016 Dec 31;6(2):226-231. doi: 10.1016/j.molmet.2016.12.009. eCollection 2017 Feb. PMID 28180064